CLINICAL TRIAL: NCT05646381
Title: A Randomized Double-blind, Placebo-controlled, Multicenter Trial Assessing the Impact of Lipoprotein(a) Lowering With Pelacarsen (TQJ230) on the Progression of Calcific Aortic Valve Stenosis [Lp(a)FRONTIERS CAVS]
Brief Title: A Multicenter Trial Assessing the Impact of Lipoprotein(a) Lowering With Pelacarsen (TQJ230) on the Progression of Calcific Aortic Valve Stenosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTQJ230A12203
Expanded Access: NCT07000695 (Available)
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Aortic Stenosis
Keywords: Cardiovascular; Lipoprotein(a); Lp(a); Hyperlipoproteinemia(a); Calcific aortic valve stenosis; TQJ230; Pelacarsen; Aortic valve stenosis; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — pelacarsen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pelacarsen (TQJ230) 80mg (Experimental): Pelacarsen (TQJ230) 80 mg prefilled syringe injected monthly, administered subcutaneously
  Interventions: Drug: Pelacarsen (TQJ230) 80mg
- Matching placebo (Placebo Comparator): Placebo to match pelacarsen (TQJ230) prefilled syringe injected monthly, administered subcutaneously
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Pelacarsen (TQJ230) 80mg — Pelacarsen (TQJ230) 80mg
  Other Names: TQJ230
  Arms: Pelacarsen (TQJ230) 80mg
Drug: Matching placebo — Matching placebo
  Other Names: Placebo
  Arms: Matching placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of pelacarsen (TQJ230) administered subcutaneously once monthly compared to placebo in slowing the progression of calcific aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥50 to <80 years of age at Screening Part II
* Lp(a) ≥175 nmol/L at the screening visit, measured at the Central laboratory
* Mild or moderate calcific aortic valve stenosis
* At the randomization visit, participant must be optimally treated for existing CV risk factors

Exclusion Criteria:

* Severe calcific aortic valve stenosis
* Uncontrolled hypertension
* History of malignancy of any organ system
* History of hemorrhagic stroke or other major bleeding
* Platelet count ≤ LLN
* Active liver disease or hepatic dysfunction
* Significant kidney disease
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2030-03-12 (Estimated); Study Completion 2030-03-12 (Estimated)

PRIMARY OUTCOMES:
Change in peak aortic jet velocity | 36 months
  To demonstrate the superiority of pelacarsen (TQJ230) vs. placebo in slowing the progression of calcific aortic valve stenosis by evaluating the change from baseline to month 36 in peak aortic jet velocity by echocardiography
Change in aortic valve calcium score | 36 months
  To demonstrate the superiority of pelacarsen (TQJ230) vs. placebo in slowing the progression of calcific aortic valve stenosis by evaluating the change from baseline to month 36 in aortic valve calcium score by computed tomography

SECONDARY OUTCOMES:
Change in Lp(a) levels | 12 months
  To assess the effect of pelacarsen (TQJ230) vs. placebo on the reduction of Lp(a) levels from baseline to month 12
Change in fibrocalcific thickening of the aortic valve | 36 months
  To assess the effect of pelacarsen (TQJ230) vs. placebo in slowing the progression of CAVS by evaluating the change from baseline to month 36 in fibrocalcific thickening of the aortic valve by contrast CT
Time from randomization to first occurrence of composite clinical endpoint event | Up to 36 months
  To assess the effect of pelacarsen (TQJ230) vs. placebo in reducing the risk of composite clinical endpoint defined as reaching either:
  1. Unplanned CAVS related hospital admission
  2. Aortic valve intervention
  3. Death related to calcific aortic valve stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (115):
- United States (34):
  - Heart Center Research Llc, Huntsville, Alabama
  - Cardiovascular Res Found, Beverly Hills, California
  - National Heart Institute, Beverly Hills, California
  - Flourish Clinical Resrch Covin, Covina, California
  - Valley Clinical Trials, Northridge, California
  - Stanford University Medical Center, Palo Alto, California
  - University Of California San Diego, San Diego, California
  - UC San Francisco Medical Center, San Francisco, California
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Nova Clinical Research LLC, Bradenton, Florida
  - Flourish Res Acq LLC North Miami, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Advanced Research for Health Improvement LLC, Naples, Florida
  - Midwest Heart and Vascular Spec, Overland Park, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hosp Harvard Med School, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - AA Medical Research Center, Flint, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University Of Minnesota, Minneapolis, Minnesota
  - Overlook Medical Center, Summit, New Jersey
  - Capital Cardiology Associates, Albany, New York
  - New York Presbyterian Hospital, New York, New York
  - Icahn School of Med at Mt Sinai, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Lindner Ctr At The Christ Hosp, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Orion Medical, Houston, Texas
  - Virginia Heart, Falls Church, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
- Austria (3):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Genk, Limburg
  - Novartis Investigative Site, Yvoir, Namur
  - Novartis Investigative Site, Aalst, Oost Vlaanderen
  - Novartis Investigative Site, Kortrijk, West-Vlaanderen
  - Novartis Investigative Site, Roeselare, West-Vlaanderen
- Canada (5):
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, North York, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (3):
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Jaroměř
  - Novartis Investigative Site, Prague
- Denmark (4):
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Hvidovre
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Viborg
- France (4):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
- Germany (14):
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Kaiserslautern, Rhineland-Palatinate
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Ahaus
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Oldenburg
- Israel (7):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (10):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Caserta, CE
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pordenone, PN
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Nieuwegein, Utrecht
- Portugal (4):
  - Novartis Investigative Site, Alcabideche
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Vila Nova de Gaia
- Spain (5):
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Zurich
- United Kingdom (9):
  - Novartis Investigative Site, Portadown, Nothern Ireland
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Londonderry
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with the applicable laws and regulations.

REFERENCES:
- [Derived] Nicholls SJ, Nelson AJ, Michael LF. Oral agents for lowering lipoprotein(a). Curr Opin Lipidol. 2024 Dec 1;35(6):275-280. doi: 10.1097/MOL.0000000000000953. Epub 2024 Sep 25. PMID 39329200